CLINICAL TRIAL: NCT02065570
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate Higher Versus Standard Adalimumab Dosing Regimens for Induction and Maintenance Therapy in Subjects With Moderately to Severely Active Crohn's Disease and Evidence of Mucosal Ulceration
Brief Title: Study to Evaluate Efficacy and Safety of Two Drug Regimens in Subjects With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-115; 2013-001746-33 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Induction: Standard Induction Dose (Experimental): Participants randomized to receive received blinded adalimumab 160 mg at Baseline and matching placebo at Week 1, adalimumab 80 mg and matching placebo at Week 2, matching placebo at Week 3, and then adalimumab 40 mg every other week (eow) starting at Week 4 through Week 12.
  Interventions: Drug: Adalimumab; Drug: Placebo
- Induction: Higher Induction Dose (Experimental): Participants randomized to receive blinded adalimumab 160 mg at Baseline, Week 1, Week 2, and Week 3. At Week 4, participants receive adalimumab 40 mg eow through Week 12.
  Interventions: Drug: Adalimumab
- Maintenance: Clinically Adjusted (CA) Regimen (Experimental): Participants randomized to the CA regimen receive adalimumab 40 mg eow beginning at Week 12. The adalimumab dose will be escalated to every week (ew) starting as early as Week 14 and up to Week 54 based on Crohn's Disease Activity Index (CDAI) or high-sensitivity C-reactive protein (hs-CRP) values, using results from the prior or current study visit. Once participants in the CA regimen are escalated, they remain on adalimumab 40 mg ew dosing.
  Interventions: Drug: Adalimumab
- Maintenance: Therapeutic Drug Monitoring (TDM) Regimen (Experimental): At Weeks 14, 28 and 42, the adalimumab dose for participants randomized to the TDM will be determined by protocol-established dose adjustment criteria. Doses will be determined using blinded serum concentrations at the prior visit (Weeks 12, 26 and 40, respectively) as well as the CDAI or hs-CRP values from the current or prior study visit. Participants who meet criteria for dose escalation at Weeks 14, 28 or 42 will receive 40 mg ew.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira
Drug: Placebo
  Arms: Induction: Standard Induction Dose

SUMMARY:
This study will evaluate higher versus standard adalimumab dosing regimens for induction and maintenance therapy in subjects with moderately to severely active Crohn's Disease and evidence of mucosal ulceration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease (CD) for at least 90 days, confirmed by endoscopy during the Screening Period.
* Active CD with a Crohn's Disease Activity Index (CDAI) despite treatment with oral corticosteroids and/or immunosuppressants.
* Mucosal ulceration on endoscopy.

Exclusion Criteria:

* Subject with ulcerative colitis or indeterminate colitis.
* Subject who has had surgical bowel resections in the past 6 months or is planning resection.
* Subjects with an ostomy or ileoanal pouch.
* Subject with symptomatic bowel stricture or abdominal or peri-anal abcess.
* Subject who has short bowel syndrome.
* Chronic recurring infections or active Tuberculosis (TB).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (143):
- United States (48):
  - Birmingham Gastroenterology Associates O.C /ID# 137282, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast /ID# 122483, Dothan, Alabama
  - Moore UC San Diego Cancer Center /ID# 119053, La Jolla, California
  - Axis Clinical Trials /ID# 130390, Los Angeles, California
  - Rocky Mountain Gastroenterology /ID# 119038, Wheat Ridge, Colorado
  - Medical Research Ctr CT /ID# 119037, Hamden, Connecticut
  - Gastroenterology Group Naples /ID# 122493, Naples, Florida
  - Internal Med Specialists /ID# 137737, Orlando, Florida
  - Shafran Gastroenterology Ctr /ID# 119057, Winter Park, Florida
  - Winship Cancer Institute of Emory University /ID# 136851, Atlanta, Georgia
  - Atlanta Gastro Assoc /ID# 119065, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 119056, Macon, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 119043, Chicago, Illinois
  - University of Chicago DCAM /ID# 119077, Chicago, Illinois
  - Carle Foundation Hospital Digestive Health Research Center /ID# 136008, Urbana, Illinois
  - Louisana Research Center, LLC /ID# 136749, Shreveport, Louisiana
  - Investigative Clinical Research /ID# 119033, Annapolis, Maryland
  - MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 119042, Chevy Chase, Maryland
  - Commonwealth Clinical Studies /ID# 136850, Brockton, Massachusetts
  - University of Michigan Health Systems /ID# 119076, Ann Arbor, Michigan
  - Minnesota Gastroenterology, P. A. /ID# 137280, Plymouth, Minnesota
  - Mayo Clinic /ID# 122489, Rochester, Minnesota
  - Kansas City Research Institute /ID# 119034, Kansas City, Missouri
  - Ctr for Digest and Liver Dis /ID# 119040, Mexico, Missouri
  - Albany Medical College /ID# 140200, Albany, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 119035, Great Neck, New York
  - The Mount Sinai Hospital /ID# 127116, New York, New York
  - Charlotte Gastroenterology and Hepatology, PLLC /ID# 119041, Charlotte, North Carolina
  - Wake Research Associates, LLC /ID# 119029, Raleigh, North Carolina
  - Consultants for Clinical Res /ID# 119052, Cincinnati, Ohio
  - Gastro United of Tulsa /ID# 122485, Tulsa, Oklahoma
  - The Oregon Clinic, Gastroenterology - West /ID# 135272, Portland, Oregon
  - West Bay Clinical Research /ID# 138330, Warwick, Rhode Island
  - Medical University of South Carolina /ID# 138122, Charleston, South Carolina
  - Erlanger Institute for Clinical Research /ID# 129008, Chattanooga, Tennessee
  - Gastro One /ID# 119068, Germantown, Tennessee
  - Nashville Med Res Inst /ID# 119050, Nashville, Tennessee
  - Vanderbilt Univ Med Ctr /ID# 125501, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas /ID# 138121, Dallas, Texas
  - Baylor College of Medicine /ID# 137277, Houston, Texas
  - Austin Institute for Clinical Research /ID# 125500, Pflugerville, Texas
  - Texas Digestive Disease Consultants - Southlake /ID# 137283, Southlake, Texas
  - Advanced Research Institute /ID# 119048, Ogden, Utah
  - University of Utah /ID# 119062, Salt Lake City, Utah
  - Gastro Assoc of Tidewater /ID# 135897, Chesapeake, Virginia
  - New River Valley Research Inst /ID# 127807, Christiansburg, Virginia
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC /ID# 119036, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital /ID# 119081, Milwaukee, Wisconsin
- Austria (5):
  - KH der Elisabethinen Linz GmbH /ID# 126280, Linz, Upper Austria
  - Medizinische Universitat Wien /ID# 126279, Vienna, Vienna
  - Medizinische Universitat Innsbruck,Universitatsklinik fur Innere Medizin 1 /ID# 126249, Innsbruck
  - LKH Salzburg and Paracelsus /ID# 126248, Salzburg
  - Krankenhaus der Barmherzigen Bruder /ID# 126270, Sankt Veit an der Glan
- Belgium (5):
  - AZ Maria Middelares /ID# 126194, Ghent
  - AZ Sint-Lucas /ID# 126242, Ghent
  - UZ Leuven /ID# 126240, Leuven
  - CHU de Liege /ID# 126241, Liège
  - AZ-Delta /ID# 126195, Roeselare
- Canada (8):
  - University of Calgary Cumming School of Medicine Adult Cystic Fibrosis Clinic /ID# 119017, Calgary, Alberta
  - University of Alberta /ID# 119022, Edmonton, Alberta
  - Winnipeg Regional Health Authority /ID# 119015, Winnipeg, Manitoba
  - Qe Ii Hsc /Id# 127115, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 119024, Greater Sudbury, Ontario
  - London Health Sciences Centre - University Hospital /ID# 119026, London, Ontario
  - Toronto Digestive Disease Asso /ID# 119019, Vaughan, Ontario
  - Montreal General Hospital - McGill University Health Center /ID# 119025, Montreal, Quebec
- Czechia (5):
  - Fakultni Nemocnice Olomouc /ID# 126264, Olomouc, Olomoucký kraj
  - Nemocnice Ceske Budejovice a.s. /ID# 126266, České Budějovice
  - Hepato-Gastroenterologie HK s.r.o. /ID# 126269, Hradec Králové
  - ISCARE a.s. /ID# 137977, Prague
  - Krajska zdravotni a.s. Masarykova nemocnice v Usti nad Labem o.z. /ID# 138331, Ústí nad Labem
- Denmark (2):
  - Herlev Hospital /ID# 127741, Herlev, Capital Region
  - Silkeborg Hospital /ID# 126251, Silkeborg
- France (7):
  - CHRU Lille - Hopital Claude Huriez /ID# 127743, Lille, Hauts-de-France
  - CHU NANCY - Hopital Brabois Adultes /ID# 127742, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Amiens-Picardie Site Sud /ID# 126237, Amiens, Somme
  - Centre Hospitalier Universitaire de Grenoble - Hopital Michallon /ID# 126200, Grenoble
  - Hopital l'Archet 2 /ID# 126238, Nice
  - CHU de Saint-Etienne, Hopital Nord /ID# 134450, Saint-Etienne
  - Hopital Rangueil /ID# 126239, Toulouse
- Germany (9):
  - Universitaetsklinikum Schleswig-Holstein /ID# 126260, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin /ID# 126196, Berlin
  - Private Practice - Dr. Michael R. MroB Dipl. med. S. Schache /ID# 126257, Berlin
  - Israelitisches Krankenhaus Hamburg /ID# 136549, Hamburg
  - Asklepios Westklinikum Hamburg /ID# 126275, Hamburg
  - Universitaetsklinikum Jena /ID# 126261, Jena
  - EUGASTRO GmbH /ID# 126259, Leipzig
  - Universitatsklinikum Magdeburg /ID# 126256, Magdeburg
  - Gastro Campus Research GbR /ID# 126274, Münster
- Hungary (4):
  - Semmelweis Egyetem /ID# 137896, Budapest
  - Magyar Elhizastudomanyi KKft. /ID# 126276, Budapest
  - Pecsi Tudomanyegyetem Klinikai l.sz. Belgyogyaszati Klinika /ID# 137895, Pécs
  - University of Szeged /ID# 126263, Szeged
- Israel (4):
  - Rabin Medical Center /ID# 126198, Petakh Tikva, Tel Aviv
  - Soroka University Medical Center /ID# 126243, Beersheba
  - Gastroenterology Institute, Division of Medicine /ID# 126245, Jerusalem
  - Kaplan Medical Center /ID# 126246, Rehovot
- Italy (7):
  - UOSD - Azienda Ospedaliera San Camillo Forlanini /ID# 127745, Rome, Lazio
  - Policlinico Agostino Gemelli /ID# 127746, Rome, Lazio
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 126221, Milan, Lombardy
  - IBD Center - IRCCS Istituto Clinico Humanitas /ID# 126226, Rozzano, Milano
  - Azienda Ospedaliera Spedali Civili /ID# 127744, Brescia
  - Azienda Ospedaliera di Padova /ID# 126267, Padua
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 129856, San Giovanni Rotondo
- Netherlands (3):
  - Academisch Medical center Amsterdam /ID# 126227, Amsterdam, North Holland
  - Erasmus Medisch Centrum /ID# 126228, Rotterdam
  - Sint Franciscus Gasthuis /ID# 127877, Rotterdam
- Poland (6):
  - Endoterapia PFG sp. z o.o. /ID# 126199, Warsaw, Masovian Voivodeship
  - Centrum Endoskopii Zabiegowej /ID# 126272, Bydgoszcz
  - Centrum Medyczne sw. Lukasza Sp. z o.o. /ID# 126271, Częstochowa
  - KO-Med Centra Kliniczne Pulawi /ID# 126278, Puławy
  - NZOZ Vivamed /ID# 126255, Warsaw
  - Centrum.Medyczne. Szpital Swietej Rodziny /ID# 137974, Lodz, Łódź Voivodeship
- School of Medicine University of Puerto Rico-Medical Science Campus /ID# 137735, San Juan, Puerto Rico
- Romania (5):
  - Institutul Clinic Fundeni /ID# 127747, Sector 2, București
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL /ID# 126277, Brasov
  - Tvm Med Serv Srl /Id# 126268, Cluj-Napoca
  - Cabinet Medical Dr. Fratila SRL /ID# 126247, Oradea
  - Salvo-san Ciobanca SRL / Medicina Interna /ID# 126224, Zalău
- Slovakia (4):
  - Gastroenterologicke centrum ASSIDUO a IBD centrum /ID# 126262, Bratislava
  - Gastroenterologicka ambulancia /ID# 137964, Bratislava
  - Vseobecna Nemocnica s poliklinikou Lucenec n.o. /ID# 127748, Lučenec
  - Poliklinika Libris /ID# 126222, Nové Mesto nad Váhom
- Spain (8):
  - Hospital Parc Tauli de Sabadell /ID# 138124, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 140425, Majadahonda, Madrid
  - Hospital Clinic /ID# 127749, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 137976, Girona
  - Hospital de Leon /ID# 141675, León
  - Hospital Clinico Universitario San Carlos /ID# 126253, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 138126, Pontevedra
  - Hospital Clinico Universitario Lozano Blesa /ID# 126252, Zaragoza
- Switzerland (2):
  - Kantonsspital St. Gallen /ID# 127750, Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Zuerich /ID# 127751, Zurich, Canton of Zurich
- Ukraine (5):
  - State Institution L. T. Malaya Therapy National Institution of NAMS of Ukraine /ID# 127753, Kharkiv, Kharkivs’ka Oblast’
  - Public Institution Kherson City Clinical Hospital named after le.le. Karabelesha /ID# 127754, Kherson
  - Kyiv City Clinical Hospital No.8 /ID# 126232, Kiev
  - Lviv Regional Clinical Hospital /ID# 126234, Lviv
  - Public Institution 6th City Clinical Hospital /ID# 126236, Zaporizhzhia
- United Kingdom (5):
  - Guy's and St Thomas' NHS Found /ID# 144366, London, London, City of
  - Norfolk and Norwich Univ Hosp /ID# 126197, Norwich, Norfolk
  - Hull University Teaching Hospitals NHS Trustust /ID# 126265, Hull
  - University Hospital Southampton NHS Fundation Trust /ID# 126225, Southampton
  - The Royal Wolverhampton NHS Tr /ID# 126201, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Battat R, Kandi S, Lacerda AP, Levine P, Neimark E, Feagan BG, Rubin DT, Ji QC, Chen X, Polakow SB. Association of bile acid diarrhea with symptoms and disease activity in Crohn's disease: post-hoc clinical trial analysis of serum 7a-hydroxy-4cholestern-3-one, C4, in patients with active Crohn's disease. J Crohns Colitis. 2025 May 8;19(5):jjaf053. doi: 10.1093/ecco-jcc/jjaf053. PMID 40202488
- [Derived] Reppell M, Zheng X, Dreher I, Blaes J, Regan E, Haslberger T, Guay H, Pivorunas V, Smaoui N. HLA-DQA1*05 Associates With Anti-Tumor Necrosis Factor Immunogenicity and Low Adalimumab Trough Concentrations in Inflammatory Bowel Disease Patients From the SERENE Ulcerative Colitis and Crohn's Disease Studies. J Crohns Colitis. 2025 Jan 11;19(1):jjae129. doi: 10.1093/ecco-jcc/jjae129. PMID 39162746
- [Derived] Verstockt B, Pivorunas V, Al Mahi N, Smaoui N, Guay H, Kennedy NA, Goodhand JR, Lin S, Bai BYH, Hanauer SB, Ferrante M, Panes J, Vermeire S. Baseline TREM-1 Whole Blood Gene Expression Does Not Predict Response to Adalimumab Treatment in Patients with Ulcerative Colitis or Crohn's Disease in the SERENE Studies. J Crohns Colitis. 2024 Apr 23;18(4):493-505. doi: 10.1093/ecco-jcc/jjad170. PMID 37801628
- [Derived] Ponce-Bobadilla AV, Stodtmann S, Chen MJ, Winzenborg I, Mensing S, Blaes J, Haslberger T, Laplanche L, Dreher I, Mostafa NM. Assessing the Impact of Immunogenicity and Improving Prediction of Trough Concentrations: Population Pharmacokinetic Modeling of Adalimumab in Patients with Crohn's Disease and Ulcerative Colitis. Clin Pharmacokinet. 2023 Apr;62(4):623-634. doi: 10.1007/s40262-023-01221-x. Epub 2023 Mar 11. PMID 36905528
- [Derived] D'Haens GR, Sandborn WJ, Loftus EV Jr, Hanauer SB, Schreiber S, Peyrin-Biroulet L, Panaccione R, Panes J, Baert F, Colombel JF, Ferrante M, Louis E, Armuzzi A, Zhou Q, Goteti VS, Mostafa NM, Doan TT, Petersson J, Finney-Hayward T, Song AP, Robinson AM, Danese S. Higher vs Standard Adalimumab Induction Dosing Regimens and Two Maintenance Strategies: Randomized SERENE CD Trial Results. Gastroenterology. 2022 Jun;162(7):1876-1890. doi: 10.1053/j.gastro.2022.01.044. Epub 2022 Feb 3. PMID 35122766
- [Derived] Greener T, Boland K, Milgrom R, Ben-Bassat O, Steinhart AH, Silverberg MS, Narula N. Higher adalimumab maintenance regimen is more effective than standard dose in anti-TNF experienced Crohn's disease patients. Eur J Gastroenterol Hepatol. 2021 Oct 1;33(10):1274-1279. doi: 10.1097/MEG.0000000000002250. PMID 34402466
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 3:2 ratio at Baseline to receive a higher induction adalimumab regimen or standard induction adalimumab regimen during the double-blind Induction Study. At Week 12, participants were re-randomized in a 1:1 ratio to a double-blind exploratory treatment regimen (adalimumab clinically adjusted [CA] regimen or adalimumab therapeutic drug monitoring [TDM] regimen).
Groups:
- Maintenance: Clinically Adjusted (CA) Regimen: Participants randomized to the CA regimen receive adalimumab 40 mg eow beginning at Week 12. The adalimumab dose could be escalated to every week (ew) starting as early as Week 14 and up to Week 54 based on Crohn's Disease Activity Index (CDAI) or high-sensitivity C-reactive protein (hs-CRP) values, using results from the prior or current study visit. Once participants in the CA regimen are escalated, they remain on adalimumab 40 mg ew dosing.
- Maintenance: Therapeutic Drug Monitoring (TDM) Regimen: At Weeks 14, 28 and 42, the adalimumab dose for participants randomized to the TDM are determined by protocol-established dose adjustment criteria. Doses are determined using blinded serum concentrations at the prior visit (Weeks 12, 26 and 40, respectively) as well as the CDAI or hs-CRP values from the current or prior study visit. Participants who meet criteria for dose escalation at Weeks 14, 28 or 42 receive 40 mg ew.
Period: Induction Study
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose | Maintenance: Clinically Adjusted (CA) Regimen | Maintenance: Therapeutic Drug Monitoring (TDM) Regimen
Started | 206 | 308 | 0 | 0
Completed | 192 | 287 | 0 | 0
Not Completed | 14 | 21 | 0 | 0
Not completed — Adverse Event | 5 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Other, Not Specified | 6 | 5 | 0 | 0
Period: Maintenance Study
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose | Maintenance: Clinically Adjusted (CA) Regimen | Maintenance: Therapeutic Drug Monitoring (TDM) Regimen
Started | 0 | 0 | 109 | 109
Completed | 0 | 0 | 87 | 90
Not Completed | 0 | 0 | 22 | 19
Not completed — Adverse Event | 0 | 0 | 8 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Other, Not Specified | 0 | 0 | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose | Total
Number analyzed (Participants) | 206 | 308 | 514
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.79) | 36.4 (13.02) | 36.4 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 158 | 267
  Male | 97 | 150 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 201 | 298 | 499
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 11 | 29
  White | 182 | 288 | 470
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 4
Description: Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 4
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Induction: Standard Induction Dose: Participants randomized to receive received blinded adalimumab 160 mg at Baseline and matching placebo at Week 1, adalimumab 80 mg and matching placebo at Week 2, matching placebo at Week 3, and then adalimumab 40 mg eow starting at Week 4 through Week 12.
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 43.7 | 43.5
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.939, Cochran-Mantel-Haenszel — Adjusted for previous infliximab use (or prior anti-tumor necrosis factor (TNF) use for participants randomized under original protocol), hs-CRP at Baseline (<10 mg/L, >=10 mg/L) and Crohn's disease severity at Baseline (CDAI ≤ 300, CDAI > 300); Adjusted risk difference = 0.3, 95% CI 2-sided [-8.1 to 8.8] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

2. Primary Outcome: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response was scored using the Simplified Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease. Endoscopic response was defined as SES-CD total score > 50% from Baseline (or for a Baseline SES-CD of 4, at least a 2 point reduction from Baseline) at Week 12.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 39.3 | 42.9
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.462, Cochran-Mantel-Haenszel — Adjusted for previous infliximab use (or prior anti-TNF use for participants randomized under original protocol), hs-CRP at Baseline (<10 mg/L, >=10 mg/L) and Crohn's disease severity at Baseline (CDAI ≤ 300, CDAI > 300); Adjusted risk difference = 3.2, 95% CI 2-sided [-5.3 to 11.7] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE): any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. Serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. TEAEs: any event that began or worsened in severity after the first dose of study drug in the induction or maintenance study. Events with unknown severity were counted as severe. Events with unknown relationship to study drug were counted as drug-related.
Time Frame: From first dose of study drug until 70 days following last dose of study drug in the induction study (up to 12 weeks) or maintenance study (up to 56 weeks).
Population: Safety Set: all participants who received at least one injection of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Induction: Standard Induction Dose: Participants were randomized to receive received blinded adalimumab 160 mg at Baseline and matching placebo at Week 1, adalimumab 80 mg and matching placebo at Week 2, and then matching placebo at Week 3, and then adalimumab 40 mg every other week (eow) starting at Week 4 through Week 12.
- Maintenance: Clinically Adjusted (CA) Regimen: Participants randomized to the CA regimen receive adalimumab 40 mg eow beginning at Week 12. The adalimumab dose will be escalated to ew starting as early as Week 14 and up to Week 54 based on CDAI or hs-CRP values, using results from the prior or current study visit. Once participants in the CA regimen are escalated, they remain on adalimumab 40 mg ew dosing.
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose | Maintenance: Clinically Adjusted (CA) Regimen | Maintenance: Therapeutic Drug Monitoring (TDM) Regimen
Number analyzed (Participants) | 206 | 308 | 109 | 109
Participants
  Any TEAE | 133 | 185 | 77 | 76
  TEAE w/reasonable possibility of being related to study drug | 54 | 75 | 29 | 33
  Any severe TEAE | 13 | 17 | 7 | 6
  Any SAE | 10 | 14 | 5 | 7
  Any TEAE leading to discontinuation of study drug | 8 | 13 | 8 | 9
  Any TEAE leading to death | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Sustained Clinical Remission (Per CDAI) at Both Weeks 4 and 12
Description: CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 4 and Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 35.0 | 39.0
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.269, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 4.6, 95% CI 2-sided [-3.6 to 12.8] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

5. Secondary Outcome: Percentage of Participants Who Achieve Clinical Response at Week 4 and Endoscopic Response at Week 12
Description: Clinical response was scored using CDAI, which assesses the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450. Clinical response was defined as a decrease in CDAI ≥ 70 points from Baseline.
  Endoscopic response was scored using the SES-CD, which evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy. The total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease. Endoscopic response was defined as SES-CD total score >50% from Baseline (or for Baseline SES-CD of 4, at least a 2-point reduction from Baseline) at Week 12.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 20.4 | 22.1
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.610, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 1.8, 95% CI 2-sided [-5.1 to 8.7] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

6. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 12
Description: Clinical remission was scored using the CDAI. CDAI assesses the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 51.5 | 62.3
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 11.2, 95% CI 2-sided [2.9 to 19.6] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

7. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use and Achieved Clinical Remission at Week 12 Among Participants Taking Corticosteroids at Baseline
Description: as for outcome 6
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Participants taking corticosteroids at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 100 | 155
percentage of participants | 48.0 | 52.9
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.336, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 6.0, 95% CI 2-sided [-6.2 to 18.2] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

8. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission was scored using the SES-CD.The SES-CD evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease. Endoscopic remission was defined as SES-CD ≤ 4 and at least a 2-point reduction versus baseline and no subscore greater than 1 in any individual variable.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 26.2 | 28.6
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.694, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 1.5, 95% CI 2-sided [-6.1 to 9.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

9. Secondary Outcome: Change From Baseline in Fecal Calprotectin Level at Week 4
Time Frame: Baseline, Week 4
Population: Intent to Treat Population: all participants who were randomized. Participants with a baseline and Week 4 assessment. Observed cases.
Measure: Mean (Standard Deviation); unit: µg/g
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 152 | 252
µg/g | -1045.7 (1648.51) | -1157.0 (2000.69)
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.946, Cochran-Mantel-Haenszel; LS Mean of Difference = 6.8, 95% CI 2-sided [-192.3 to 205.9]

10. Secondary Outcome: Percentage of Participants With Hs-CRP < 5 mg/L and Fecal Calprotectin < 250 µg/g at Week 4
Time Frame: Week 4
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 27.7 | 32.5
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.293, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 4.0, 95% CI 2-sided [-3.5 to 11.5] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

11. Secondary Outcome: Percentage of Participants With Clinical Remission, Hs-CRP < 5 mg/L and Fecal Calprotectin < 250 µg/g at Week 4
Description: as for outcome 6
Time Frame: Week 4
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 11.2 | 14.3
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 3.0, 95% CI 2-sided [-2.7 to 8.6] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

12. Secondary Outcome: Percentage of Participants With Clinical Remission, Hs-CRP < 5 mg/L and Fecal Calprotectin < 250 µg/g and Endoscopic Remission at Week 12
Description: Clinical remission was scored using the CDAI. CDAI assesses the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
  Endoscopic remission was scored using the SES-CD.The SES-CD evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy. The total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease. Endoscopic remission was defined as SES-CD ≤ 4 and at least a 2-point reduction versus baseline and no subscore greater than 1 in any individual variable.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 7.3 | 11.7
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.092, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 4.2, 95% CI 2-sided [-0.7 to 9.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

13. Secondary Outcome: Percentage of Participants Who Achieved an SES-CD ≤ 2 at Week 12
Description: The SES-CD evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 16.0 | 20.1
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.278, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 3.6, 95% CI 2-sided [-2.9 to 10.2] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

14. Secondary Outcome: Percentage of Participants With Clinical Response at Week 4
Description: Clinical response was scored using CDAI is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450. Clinical response was defined as a decrease in CDAI ≥ 70 points from baseline.
Time Frame: Week 4
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 70.9 | 74.4
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.353, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 3.7, 95% CI 2-sided [-4.1 to 11.5] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

15. Secondary Outcome: Percentage of Participants With Clinical Response at Week 12
Description: Clinical response was scored using CDAI. CDAI assesses the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450. Clinical response was defined as a decrease in CDAI ≥ 70 points from Baseline.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 74.8 | 83.4
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 8.9, 95% CI 2-sided [1.8 to 16.0] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

16. Secondary Outcome: Percentage of Participants Achieving Response in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Symptom Domain at Week 4
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). The range for Bowel Symptom domain score is 10 (severe problem) to 70 (normal health). Response in IBDQ Bowel Symptom domain is defined as an increase of IBDQ Bowel Symptom domain score ≥ 8.
Time Frame: Week 4
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 71.4 | 74.7
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.394, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 3.4, 95% CI 2-sided [-4.4 to 11.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

17. Secondary Outcome: Percentage of Participants Achieving Response in IBDQ Bowel Symptom Domain at Week 12
Description: as for outcome 16
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 73.3 | 76.9
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.349, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 3.6, 95% CI 2-sided [-4.0 to 11.2] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

18. Secondary Outcome: Percentage of Participants Achieving Response in IBDQ Fatigue Item at Week 12
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). The IBDQ Fatigue item score range is from 1 (severe problem) to 7 (normal health). Response is defined as an increase of IBDQ Fatigue item score ≥ 1.
Time Frame: Week 12
Population: Intent to Treat Population: all participants who were randomized. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose
Number analyzed (Participants) | 206 | 308
percentage of participants | 68.4 | 76.0
Statistical Analysis 1: Comparison: Induction: Standard Induction Dose vs Induction: Higher Induction Dose; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted risk difference = 7.6, 95% CI 2-sided [-0.1 to 15.3] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 70 days following last dose of study drug in the induction study (up to 12 weeks) or maintenance study (up to 56 weeks).
Groups:
- Maintenance: Therapeutic Drug Management (TDM) Regimen: At Weeks 14, 28 and 42, the adalimumab dose for participants randomized to the TDM are determined by protocol-established dose adjustment criteria. Doses are determined using blinded serum concentrations at the prior visit (Weeks 12, 26 and 40, respectively) as well as the CDAI or hs-CRP values from the current or prior study visit. Participants who meet criteria for dose escalation at Weeks 14, 28 or 42 receive 40 mg ew.
Arm/Group | Induction: Standard Induction Dose | Induction: Higher Induction Dose | Maintenance: Clinically Adjusted (CA) Regimen | Maintenance: Therapeutic Drug Management (TDM) Regimen
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/308 | 0/109 | 0/109
Serious Adverse Events (participants affected / at risk) | 10/206 | 14/308 | 5/109 | 7/109
Other Adverse Events (participants affected / at risk) | 54/206 | 58/308 | 41/109 | 33/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Standard Induction Dose (N=206) | Induction: Higher Induction Dose (N=308) | Maintenance: Clinically Adjusted (CA) Regimen (N=109) | Maintenance: Therapeutic Drug Management (TDM) Regimen (N=109)
SCLERITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACQUIRED IMMUNODEFICIENCY SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VARICELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAPILLARY RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SELECTIVE ABORTION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Standard Induction Dose (N=206) | Induction: Higher Induction Dose (N=308) | Maintenance: Clinically Adjusted (CA) Regimen (N=109) | Maintenance: Therapeutic Drug Management (TDM) Regimen (N=109)
CROHN'S DISEASE (Gastrointestinal disorders) | 12 (14) | 14 (15) | 16 (20) | 15 (17)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (7) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 15 (17) | 9 (10) | 5 (7) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 9 (11) | 19 (21) | 15 (15) | 10 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 (19) | 10 (10) | 8 (8) | 4 (5)
DIZZINESS (Nervous system disorders) | 11 (13) | 2 (2) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 18 (24) | 17 (19) | 9 (9) | 8 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02065570/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02065570/SAP_001.pdf